CLINICAL TRIAL: NCT03320239
Title: Using HIV Risk Assessment Tool to Promote HIV Testing Among Men Who Have Sex With Men in Beijing: a Social Media-based Randomized Trial
Brief Title: Using HIV Risk Assessment Tool to Promote HIV Testing Among Men Who Have Sex With Men
Acronym: online-RASSL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: risk assessment
Record Dates: First submitted 2017-10-17; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: HIV/AIDS; HIV Infections; Social Media
Keywords: HIV; risk assessment; HIV testing; unprotected anal intercourse; Social medica
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the online-RASSL intervention group (Experimental): HIV risk assessment and tailored suggestions, free HIV testing link
  Interventions: Behavioral: HIV risk assessment and tailored suggestions
- intervention group 2 (Experimental): HIV risk behavior investigation and routine education
  Interventions: Behavioral: HIV risk behavior assessment
- the control group (Placebo Comparator): The placebo control: HIV/AIDS knowledge assessment, routine education
  Interventions: Behavioral: placebo control

INTERVENTIONS:
Behavioral: HIV risk assessment and tailored suggestions — The intervention contains: HIV risk investigation, tailored suggestions and free HIV testing link
  Arms: the online-RASSL intervention group
Behavioral: HIV risk behavior assessment — It only contains HIV risk behavior assessment and routine education
  Arms: intervention group 2
Behavioral: placebo control — It only contains HIV/AIDS knowledge assessment and routine education
  Arms: the control group

SUMMARY:
The objective of the study is to evaluate the effectiveness of a HIV risk assessment tool to promote HIV testing and to reduce high risk sexual behaviors among men who have sex with men (MSM). It hypothesizes that the social media-based HIV risk assessment tool can increase 20% HIV testing proportion during the six months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male at birth.
* Having had homo-sexual behaviors (anal/oral) in the past 6 months before enrollment.
* An age of 18 years or older.
* Living in Beijing, China.
* Self-reporting HIV negative or unknown.
* Willingly participating into the baseline survey and the six months follow ups.
* Agreeing not to share the research link to others.
* Owning a mobile phone and having had downloaded the social networking Application Blued before enrollment.

Exclusion Criteria:

* Not accepting blood sampling within the study period.
* Reporting injecting drugs use in the past six months before enrollment.
* Being currently involved in other HIV behavioral interventions for MSM.
* Having a specific plan to leave from Beijing in the next 6 months.
* Self-reporting female.
* Other reasons the investigators deem make participation either detrimental to the participants or the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of HIV testing during the study period | 1 month
  The numerator is the number of participants who come to the specific HIV testing clinics for HIV test during the study period, the denominator is the number of participants randomized per group.

SECONDARY OUTCOMES:
unprotected anal intercourse | 6 months
  Questionaire will be used to collect the frequency of unprotected anal intercourse at month 1, month 3 and month 6 after the study starts.
Post exposure prophylaxis (PEP) | 6 months
  Questionaire will be used to collect data on whether participants use PEP at month 1, month 3 and month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Z You, PhD, Study Director — NATIONAL CENTER FOR HIV/STD CONTROL AND PREVENTION
Locations (1):
- national center for AIDS control and prevention, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Luo Q, Wu Z, Mi G, Xu J, Scott SR. Using HIV Risk Self-Assessment Tools to Increase HIV Testing in Men Who Have Sex With Men in Beijing, China: App-Based Randomized Controlled Trial. J Med Internet Res. 2023 Sep 1;25:e45262. doi: 10.2196/45262. PMID 37656500